CLINICAL TRIAL: NCT00357357
Title: Clinical Safety/Tolerability of HF0220 and Its Effect on Biochemical Markers Relevant to Patients With a Diagnosis of Mild to Moderate Alzheimer' Disease
Brief Title: European Study of HF0220 in Mild to Moderate Alzheimer's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunter-Fleming Ltd (Industry)
Responsible Party: Dr John Fox ,Chief Operations Officer, Hunter-Fleming Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HF0220/003; 2005-005791-32
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group1 (Placebo Comparator): 4x 7 day rising dose
  Interventions: Drug: HF0220
- Group2 (Placebo Comparator): 4x, 7 day rising dose
  Interventions: Drug: HF0220
- Group3 (Placebo Comparator): 28 day fixed lower dose
  Interventions: Drug: HF0220
- Group4 (Placebo Comparator): 28 day fixed upper dose
  Interventions: Drug: HF0220

INTERVENTIONS:
Drug: HF0220 — comparison of different dosages of drug

SUMMARY:
The purpose of this Phase II study is to evaluate the safety and tolerability of HF 0220 in patients with Alzheimer's disease compared to placebo (inactive substance). The study will also validate biochemical markers as appropriate clinical end-points and to assess the suitability of chosen dose levels for future clinical studies.

ELIGIBILITY:
RECRUITMENT OF PARTICIPANTS IS PERFORMED ONLY BY STUDY SITES

INCLUSION CRITERIA:

Participants must meet the following inclusion criteria to be eligible.

* Male or Female (age over 55 years). Females must be non-child-bearing potential. Male patients with female partners of child-bearing potential should use effective contraception for the duration of the Study.
* A diagnosis of probable Alzheimer's disease established in accordance with the National Institute of Neurological and Communicative Disorders and Stroke /Alzheimer's disease and Related Disorders Association (NINCDS-ADRDA) classification.
* Severity of dementia of mild to moderate as assessed by the Mini-Mental State Examination (MMSE) score of 12-24.
* Patients must be living in the community living with or have at least daily visits from a responsible carer. The carer should be capable of assisting with the patient's medication, and prepared to attend with the patient for assessment.
* Written consent should be obtained from the patient and responsible carer.

EXCLUSION CRITERIA

Patients will not be eligible to participate in the study if they meet any of the following criteria:

* Primary, secondary or pseudodementias other than probable Alzheimer's disease.
* Clinically significant and/or uncontrolled condition or other significant medical disease.
* If taking medication for symptoms of dementia, the patient must be stable on therapy and have been taking these for a minimum of 3 months prior to enrolment.
* Treatment within the previous 3 months with any drug known to have a well defined potential for hepatotoxicity.
* Non-steroidal or steroidal anti-inflammatory agents. However, patients stable on low dose aspirin (upto 300mg/day) for at least 3 month prior to enrolment will be eligible.
* Taking anti-oxidant supplements.
* Active smokers of tobacco.
* Considered to be malnourished (body mass index <19).
* Patients in whom a lumbar puncture is contra-indicated.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of HF 0220 in mild to moderate Alzheimer's patients | June 2008

SECONDARY OUTCOMES:
Validate biochemical markers relevant to Alzheimer's disease | June 2008
Assess the suitability of chosen HF0220 dose levels for future studies | June 2008

CONTACTS AND LOCATIONS:
Overall Officials: David Wilkinson, Principal Investigator — Chief Principal Investigator; Niels Andreasen, Dr, Principal Investigator — Swedish Co-Ordinating Principal Investigator
Locations (10):
- India (5):
  - King George Hospital, Visakhapatnam, ANDH PRAD
  - Manipal Hospital,, Bangalore, Karna
  - Sree Chitra Tirunal Institute for Medical Sciences and Technology, Thiruvananthapuram, Kerala
  - Nizam's Institute of Medical Sciences,, Hyderabaad, Panjagutta
  - Madras Medical College & Government General Hospital, Chennai, Tamil Nadu
- Sweden (2):
  - Malmo University Hospital, Malmo
  - Karolinksa Institute, Stockholm
- United Kingdom (3):
  - Research Institute for Care of the Elderly, Bath
  - Memory Assessment and Research Centre, Southampton
  - Kingshill Research Centre, Swindon

REFERENCES:
- [Background] Pringle AK, Schmidt W, Deans JK, Wulfert E, Reymann KG, Sundstrom LE. 7-Hydroxylated epiandrosterone (7-OH-EPIA) reduces ischaemia-induced neuronal damage both in vivo and in vitro. Eur J Neurosci. 2003 Jul;18(1):117-24. doi: 10.1046/j.1460-9568.2003.02734.x. PMID 12859344